CLINICAL TRIAL: NCT06787794
Title: The Effectiveness of Virtual Reality-assisted Hypnosis in Reducing Itch: a Proof-of-concept Study
Brief Title: Reducing Itch With Hypnosis and Virtual Reality
Acronym: VRITCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Leiden (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Antoinette van Laarhoven, Principal Investigator, Universiteit Leiden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL83542.058.23
Record Dates: First submitted 2025-01-07; First posted 2025-01-22 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: ITCH; Pruritus
Keywords: Chronic Pruritus; Chronic Itch; Therapy resistant; Virtual Reality (VR); Hypnosis; Relaxation; Distraction
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Intervention Model Description: The participants are randomised over an interventional condition and a waiting list. In case of proven effectivity, the people on the waiting list will be able to also participate at a later instance in the intervention, which will not be part of the analyses within this study.
Masking Description: No blinding possible in the current design (waiting list control)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality-assisted hypnosis (VRH) (Experimental): Participants on the VRH intervention group will come for a total of 8 sessions, including a baseline session, 6 interventional sessions, and a follow-up session.
  During the intervention period, participants are requested to perform guided self hypnosis at home according to audio fragments provided (ca. 5 min/day).
  Interventions: Behavioral: Virtual Reality-assisted hypnosis
- Waiting list control (No Intervention): Participants in the waiting list control will participate in the baseline session, final session, and follow-up session (questionnaires and cowhage application) and answer questionnaires online, weekly between baseline and the final session.

INTERVENTIONS:
Behavioral: Virtual Reality-assisted hypnosis — The VRH intervention consists of 6 interventional sessions. Every session, first, participants receive hypnotic induction and go through a deepening phase using a hypnotic script and a VR environment designed based on input from individuals suffering from chronic itch. To this end, participants are instructed to close their eyes while they will continue to listen to the recorded hypnotic script developed based on general hypnotic principles as amongst others described by Yapko (2013). Direct antipruritic suggestions are used such as "your skin will feel so soft, relaxed and cool, it is fully at ease". After these standardized suggestions, the participants will be alerted again. Home exercises (ca 5 min/day) include guided self-hypnosis records with direct antipruritic suggestions comparable to the ones they listen to during the intervention at location.
  Arms: Virtual Reality-assisted hypnosis (VRH)

SUMMARY:
Chronic itch is a disabling condition with currently limited treatment options. Virtual reality (VR) is a relatively new approach that provides immersion in another environment and has been shown to have a temporary itch mitigating potential. Hypnosis, which is a state of relaxation, has been successfully applied with more long-term treatment effects in the specific case of itch as a result of severe atopic dermatitis. However, hypnosis tends to depend on an individual's susceptibility, or ease, to come into a hypnotic state. A combination of VR and hypnosis (VRH) has been put forward since it may combine the longer lasting effects of hypnosis with VR making the hypnosis more accessible by facilitating imagination. Even though VRH is a promising avenue, it has never been investigated in the context of itch. In this randomized controlled trial, comparing a VRH treatment with a waiting list control group after 6 sessions and at follow-up, it is aimed to assess the effectiveness of VRH in reducing itch along with its psychological burden in adult individuals with therapy-resistant disabling itch.

DETAILED DESCRIPTION:
Rationale: Chronic itch is a disabling condition with currently limited treatment options. Virtual reality (VR) is a relatively new approach that provides immersion in another environment and has been shown to have a temporary itch mitigating potential. Hypnosis, which is a state of relaxation, has been successfully applied with more long-term treatment effects in the specific case of itch as a result of severe atopic dermatitis. However, hypnosis tends to depend on an individual's susceptibility, or ease to come into a hypnotic state. A combination of VR and hypnosis (VRH) has been put forward since it may combine the longer lasting effects of hypnosis with VR making the hypnosis more accessible by facilitating imagination. Even though VRH is a promising avenue, it has never been investigated in the context of itch.

Objective: This study aims to assess the effectiveness of VRH in reducing itch along with its psychological burden in individuals with chronic itch.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be adults (aged 18-80 years)
* Participants must have been suffering from chronic pruritus of any origin for at least 1 year prior to inclusion in this study
* Participants must have been seen by a physician for the itch
* Participants must experience psychological and/or functional impairment due to the itch despite standard medical treatment.
* Participants must speak and understand Dutch and be able to complete questionnaires.

Exclusion Criteria:

* Severe psychiatric comorbidities irrelated to their itch condition such as psychosis or severe clinical depression or anxiety disorder (anxiety and depressive symptoms in itself are common in individuals with chronic symptoms and therefore no reason for exclusion);
* History of seizures;
* History of severe migraine;
* Severe susceptibility to motion sickness;
* Balance problems;
* Face, head, or neck injury;
* Visual or audiological impairment;
* Pacemaker, defibrillator and/or other electronic (implantable) device of vital importance;
* Pregnancy;
* Lactation;
* Participation in another interventional itch study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical itch intensity | Baseline, immediately after the intervention, and at follow-up (±6 weeks after end of intervention)
  The primary outcome is short-term (end of treatment) and longer-term (approximately 6 weeks post-treatment) itch reduction (0-10 NRS) [end of treatment and follow-up compared to baseline; between group].

SECONDARY OUTCOMES:
Impact of Skin Disease on Daily Life (ISDL) Questionnaire | Baseline, immediately after the intervention, and at follow-up (±6 weeks after end of intervention)
  The impact of the itch on the participants' overall wellbeing is measured by the Impact of Skin Disease on Daily Life (ISDL) Questionnaire [Evers et al., 2008]. The following subscales are used: (1) skin status (items 7 t/m 10), (2) physical symptoms (items 11 to 16), (3) scratching (items 17 to 23), (4) impact of disease on daily life (items 24 and 26), (5) psychological functioning (items 27 and 28), and (6) illness cognitions (items 31 and 32).
Hospital Anxiety and Depression Scale (HADS) questionnaire | Baseline, immediately after the intervention, and at follow-up (±6 weeks after end of intervention)
  The validated HADS measuring anxiety and depression.
Medical treatment need | Baseline, during the intervention, immediately after the intervention, and at follow-up (±6 weeks after end of intervention)
  Medical treatment need defined by type of drug/treatment x quantification
itch sensitivity (to the cowhage plant particles). | Baseline, immediately after the intervention, and at follow-up (±6 weeks after end of intervention)
  25 cowhage plant particles are rubbed on the participants' forearm (or at the closest non-lesional site) for 45 seconds and the participants are asked to rate the subsequent itch sensitivity on the 0-10 NRS for itch every half minute for in total up to 4 minutes [e.g. Blythe et al., 2021; Weng et al., 2022]. Peak and average itch over the 4 minutes is being calculated.

OTHER OUTCOMES:
Clinical itch intensity | Baseline, during the intervention, immediately after the intervention, and at follow-up (±6 weeks after end of intervention)
  Akin the primary outcome, but now explored over the sessions
VRH and VR-adjusted version of the GAMQ General Attitude towards Medication Questionnaire | Baseline (in relation to treatment outcomes)
  The validated GAMQ General Attitude towards Medication Questionnaire, adjusted to the current intervention (elements) will be adminstered at baseline
Hypnotic susceptibility | Baseline (in relation to treatment outcomes)
  The validated Stanford Hypnotic Susceptibility Scale C [e.g. Näring et al., 2001]) is administered by an experienced hypnotherapist who will bring the participants in hypnosis and give the suggestions according to this scale.

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette I.M. van Laarhoven, PhD, Principal Investigator — Leiden University, Health Medical and Neuropsychology Unit
Locations (1):
- Leiden University, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data are available upon reasonable request via an online repository. As online repository, we intend to use DataverseNL, which offers a reliable and secure infrastructure. The Faculty's data stewards are in charge of uploading the publication package to DataverseNL. Files uploaded include the research protocols and outcome data (special care is taken that the information does not allow tracing to the individual patient).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Upon publication of the findings in a scientific journal - no end date
Access Criteria: Data obtained through this study may be provided to qualified researchers with academic interest in chronic itch, while detailing specific plans in relation to the data. Data shared will be anonymized. Approval of the request and execution of all applicable agreements (i.e. a Data Sharing Agreement, requiring the signature of your university's legal team) are prerequisites to the sharing of data with the requesting party. For more information, please contact datastewards_psy_ped@fsw.leidenuniv.nl.

REFERENCES:
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Weng L, van Laarhoven AIM, Peerdeman KJ, Evers AWM. Induction and generalization of nocebo effects on itch. Exp Dermatol. 2022 Jun;31(6):878-889. doi: 10.1111/exd.14522. Epub 2022 Feb 6. PMID 35000228
- [Background] Evers AW, Duller P, van de Kerkhof PC, van der Valk PG, de Jong EM, Gerritsen MJ, Otero E, Verhoeven EW, Verhaak CM, Kraaimaat FW. The Impact of Chronic Skin Disease on Daily Life (ISDL): a generic and dermatology-specific health instrument. Br J Dermatol. 2008 Jan;158(1):101-8. doi: 10.1111/j.1365-2133.2007.08296.x. Epub 2007 Nov 10. PMID 17999699
- [Background] Naring GW, Roelofs K, Hoogduin KA. The Stanford Hypnotic Susceptibility Scale, Form C: normative data of a Dutch student sample. Int J Clin Exp Hypn. 2001 Apr;49(2):139-45. doi: 10.1080/00207140108410064. PMID 11294117
- See also: Yapko, M. D. (2013). Essentials of hypnosis. Routledge. (ISBN 9781138814288) — https://www.routledge.com/Essentials-of-Hypnosis/Yapko/p/book/9781138814288?srsltid=AfmBOop8aIFv_G0Dh-Py4IR4vjAxC98aNbGd225UCZ5T02reoAzNu7Zw